CLINICAL TRIAL: NCT00283933
Title: A Phase 2, Open-Label, Single Dose Level, 24-Week Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of AT1001 in Patients With Fabry Disease
Brief Title: A 24-Week Safety and Pharmacodynamic Study of AT1001 (Migalastat Hydrochloride) in Participants With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAB-CL-203 (AA1565522)
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-08

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; AT1001; Galafold; Migalastat; Substrate
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Migalastat (Experimental): Migalastat 150 milligrams (mg) was administered orally QOD during the 24-week treatment period and then during the optional 24-week extension period.
  Interventions: Drug: migalastat HCl

INTERVENTIONS:
Drug: migalastat HCl
  Other Names: AT1001; Galafold; migalastat

SUMMARY:
Study to evaluate the safety, tolerability, and pharmacodynamics of migalastat hydrochloride (HCl) (migalastat) in participants with Fabry disease.

DETAILED DESCRIPTION:
This was a Phase 2, open-label study in male participants with Fabry disease. The study consisted of a 4-week screening period, during which participants' galactosidase (GLA) genotype was assessed for α-galactosidase A (α-Gal A) activity in response to migalastat. Participants were required to have α-Gal A activity responsive to migalastat. The study consisted of a 24-week treatment period, followed by an optional 24-week extension period. Participants received migalastat once every other day (QOD) for 24 weeks during the treatment period and the optional 24-week extension for a total treatment duration of up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 65 years of age (inclusive)
* Hemizygous for Fabry disease
* Had a confirmed diagnosis of Fabry disease with a documented missense gene mutation (individual or familial)
* Had enhanceable enzyme activity based on in vitro tests
* Had documented evidence of cardiac and/or renal dysfunction (for example, abnormal electrocardiogram (ECG), left ventricular hypertrophy, renal insufficiency)
* Were previously untreated by enzyme replacement therapy (ERT) or substrate depletion for Fabry disease, or if ERT or other specific treatment for Fabry disease was administered, were able to stop ERT for at least 30 weeks.
* Were willing to undergo 2 kidney and 3 skin biopsies
* Agreed to be sexually abstinent or use a condom with spermicide when engaging in sexual activity during the course of the study and for a period of 30 days following completion of the study
* Were willing and able to sign an informed consent form

Exclusion Criteria:

* History of significant disease other than Fabry disease (for example, end-stage renal disease; Class III or IV heart disease [per the New York Heart Association classification]; current diagnosis of cancer, except for basal cell carcinoma of the skin; diabetes [unless hemoglobin A1c ≤8]; or neurological disease that would have impaired the participant's ability to participate in the study)
* History of organ transplant
* Serum creatinine >176 millimole per deciliter on Day -2
* Screening 12-lead ECG demonstrating corrected QT interval >450 milliseconds prior to dosing
* Taking a medication prohibited by the protocol: Fabrazyme® (agalsidase beta), Replagal™ (agalsidase alfa), Glyset® (miglitol), Zavesca® (miglustat), or any experimental therapy for any indication
* Participated in a previous clinical trial in the last 30 days
* Any other condition, which, in the opinion of the investigator, would jeopardize the safety of the participant or impact the validity of the study results

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-05-09 (Actual); Primary Completion 2008-03-12 (Actual); Study Completion 2008-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (2):
- Paris, France
- London, United Kingdom

REFERENCES:
- [Derived] Benjamin ER, Della Valle MC, Wu X, Katz E, Pruthi F, Bond S, Bronfin B, Williams H, Yu J, Bichet DG, Germain DP, Giugliani R, Hughes D, Schiffmann R, Wilcox WR, Desnick RJ, Kirk J, Barth J, Barlow C, Valenzano KJ, Castelli J, Lockhart DJ. The validation of pharmacogenetics for the identification of Fabry patients to be treated with migalastat. Genet Med. 2017 Apr;19(4):430-438. doi: 10.1038/gim.2016.122. Epub 2016 Sep 22. PMID 27657681
- [Derived] Germain DP, Giugliani R, Hughes DA, Mehta A, Nicholls K, Barisoni L, Jennette CJ, Bragat A, Castelli J, Sitaraman S, Lockhart DJ, Boudes PF. Safety and pharmacodynamic effects of a pharmacological chaperone on alpha-galactosidase A activity and globotriaosylceramide clearance in Fabry disease: report from two phase 2 clinical studies. Orphanet J Rare Dis. 2012 Nov 24;7:91. doi: 10.1186/1750-1172-7-91. PMID 23176611

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period
Arm/Group | Migalastat
Started | 5
Safety Population (Received at least 1 dose of study drug) | 5
Pharmacodynamic (PD) Population (Received study drug and had at least 1 non-missing postbaseline PD parameter recorded) | 5
Completed | 5
Not Completed | 0
Period: Extension Period
Arm/Group | Migalastat
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least 1 dose of study drug.
Groups:
- Migalastat: Migalastat 150 mg was administered orally QOD during the 24-week treatment period and then during the optional 24-week extension period.
Arm/Group | Migalastat
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse event with start date on or after administration of study drug or pre-existing conditions that worsened on or after the start of the first study drug administration (on Day 1). A severe adverse event was defined as an adverse event that was incapacitating and required medical intervention. The number of participants who experienced one or more severe TEAEs after dosing on Day 1 through Week 48 is presented. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through Week 48
Population: Safety Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: α-Galactosidase A (α-Gal A) Activity In Peripheral Blood Mononuclear Cells (PBMC) At Baseline, Week 24, And Week 48
Description: PBMC were isolated from whole blood and lysed, and α-Gal A activity was measured using a validated fluorometric assay, with catalysis to fluorescent 4-methylumbelliferone (4-MU) as the activity measure. The activity values obtained were normalized to protein (measured using a colorimetric assay) and reported as enzyme activity (nanomole [nmol] 4-MU/hour [hr]) per mg of protein. On Day 1 of the first visit and at every visit thereafter, the samples were collected prior to dosing with migalastat. α-Gal A activity in leukocytes are presented by individual participants.
Time Frame: Baseline, Week 24 (end of treatment period), Week 48 (end of extension period)
Population: PD Population: All participants who received at least 1 dose of study drug and had at least 1 non-missing postbaseline PD parameter recorded.
Measure: Number; unit: nmol 4-MU/hr/mg protein
Arm/Group | Migalastat
Number analyzed (Participants) | 5
nmol 4-MU/hr/mg protein
  Participant 1: Baseline: number analyzed (Participants) | 1
  Participant 1: Baseline | 0.05
  Participant 1: Week 24: number analyzed (Participants) | 1
  Participant 1: Week 24 | 0.36
  Participant 1: Week 48: number analyzed (Participants) | 1
  Participant 1: Week 48 | 0.1
  Participant 2: Baseline: number analyzed (Participants) | 1
  Participant 2: Baseline | 0.06
  Participant 2: Week 24: number analyzed (Participants) | 1
  Participant 2: Week 24 | 0.13
  Participant 2: Week 48: number analyzed (Participants) | 1
  Participant 2: Week 48 | 0.1
  Participant 3: Baseline: number analyzed (Participants) | 1
  Participant 3: Baseline | 0.14
  Participant 3: Week 24: number analyzed (Participants) | 1
  Participant 3: Week 24 | 0.3
  Participant 3: Week 48: number analyzed (Participants) | 1
  Participant 3: Week 48 | 0.33
  Participant 4: Baseline: number analyzed (Participants) | 1
  Participant 4: Baseline | 3.4
  Participant 4: Week 24: number analyzed (Participants) | 1
  Participant 4: Week 24 | 10.9
  Participant 4: Week 48: number analyzed (Participants) | 1
  Participant 4: Week 48 | 7.4
  Participant 5: Baseline: number analyzed (Participants) | 1
  Participant 5: Baseline | 0.18
  Participant 5: Week 24: number analyzed (Participants) | 1
  Participant 5: Week 24 | 1.32
  Participant 5: Week 48: number analyzed (Participants) | 1
  Participant 5: Week 48 | 0.13

ADVERSE EVENTS:
Time Frame: Day 1 after dosing through Week 48 (end of extension period)
Arm/Group | Migalastat
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (N=5)
Ventricular tachycardia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Scrotal mass (Reproductive system and breast disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can only publish the results from this trial provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review. If requested, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.